CLINICAL TRIAL: NCT06748066
Title: Development and Validation of the RISE-ACL Scale for Assessing Risk-Taking Intension and Propensity After ACL Reconstruction
Brief Title: Developing and Validating the Risk-taking Intention and Sport Engagement After ACL Reconstruction (RISE-ACL) Scale
Acronym: RISE-ACL
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Collaborators: INSERM UMR U1075 Comète GIP Cyceron, unicaen, Caen Normandie (Unknown)
Responsible Party: Principal Investigator, Joffrey DRIGNY, Maître de conférences des universités - praticien hospitalier (MCU-PH), M.D, Ph.D, University Hospital, Caen
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: RISE-ACL
Record Dates: First submitted 2024-12-18; First posted 2024-12-24 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: ACL Surgery; ACL Injuries; ACL Reconstruction
Keywords: Postoperative Care; Return to Sport; Risk-Taking; Anterior Cruciate Ligament Injuries
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Risk-Taking

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group of experts in the field of ACL reconstruction surgery and follow-up (Experimental): A group of 11 experts in the field of ACL reconstruction, each with a minimum of five years of experience and at least 100 patients managed, will collaborate to select the items to be included in the RISE-ACL scale for assessing Risk-taking Intention and Sport Engagement after ACL reconstruction.
  Interventions: Behavioral: RISE-ACL development
- ACL - reconstruction group, scale validation (Experimental): 162 patients who have undergone ACL reconstruction within the past two years and are currently in the 'Return to Sport' process, with follow-up in the sports medicine department, will complete the RISE-ACL scale for assessing Risk-taking Intention and Sport Engagement after ACL reconstruction.
  Interventions: Behavioral: RISE-ACL scale validation

INTERVENTIONS:
Behavioral: RISE-ACL development — A meeting will be organized with all expert panel members to select relevant items. Before the meeting, experts will review a literature on ACL reconstruction return to sport processes. During round 1, the chairperson will ask panel members to suggest items to be included in the scale. Items with agreement from 5 or more members will be included in round 2. In round 2, redundant items will be identified and grouped, and new items will be added based on the literature and expert experience. Selected items will be randomly ordered to create a preliminary 6-level Likert scale (0 = strongly disagree, 5 = strongly agree).
  Arms: Group of experts in the field of ACL reconstruction surgery and follow-up
Behavioral: RISE-ACL scale validation — The scale validation phase will involve 162 participants who have undergone ACL reconstruction within the past two years and are in the 'Return to Sport' process, with follow-up in the sports medicine department.
  These participants will complete the final version of the RISE-ACL Scale in addition with the ACL-RSI scale and the IKDC Subjective Knee Form.
  Validation will consist of testing face validity, construct validity, criterion validity (concurrent validity), and reliability, including internal consistency and test-retest reliability.
  Arms: ACL - reconstruction group, scale validation

SUMMARY:
Psychological factors play a critical role in recovery following anterior cruciate ligament (ACL) reconstruction. While tools such as the ACL - Return to Sport after Injury (ACL-RSI) focus on psychological readiness, emphasizing fear, hesitation, and apprehension, the opposite spectrum-overconfidence and risk-taking behaviors-remains underexplored. These behaviors can lead to premature return to high-risk activities and an increased likelihood of re-injury.

To address this gap, we propose the development and validation of the RISE-ACL scale for assessing Risk-taking Intention and Sport Engagement after ACL reconstruction. This scale will assess key factors such as patients' willingness to engage in high-impact activities, their adherence to medical guidance, and their perceived readiness to resume sports despite potential physical or psychological limitations.

The RISE-ACL Scale will complement existing tools like the ACL-RSI by focusing on overconfidence and risk-taking, offering clinicians a more balanced perspective on psychological recovery. Validation of the scale will involve testing its validity, reliability and clinical utility to ensure accurate identification of at-risk individuals.

By providing actionable insights, the RISE-ACL Scale will help enhance post-operative care, promote safer return-to-play decisions, and optimize long-term outcomes through a comprehensive assessment of psychological and behavioral factors.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have had an ACL reconstruction surgery (isolated or associated with other meniscal or ligamentary surgery)
* Patient included in the sport medicine follow-up protocole
* Patients who have provided informed consent.

Exclusion Criteria:

* Participants who are not included in the Return-to-sport process

Ages: 16 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 162 (Actual)
Dates: Start 2025-02-03 (Actual); Primary Completion 2025-07-29 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
The RISE-ACL scale for assessing Risk-taking Intention and Sport Engagement after ACL reconstruction. | One measurement during one visit at 4 to 24 months after surgery
  The RISE-ACL Scale will measure patients' risk-taking tendencies, overconfidence in their recovery, and willingness to resume sports despite physical or psychological limitations. The number and nature of the items will be defined during the development phase. The scale will be scored on a Likert scale ranging from 0 to 3, with 0 representing "strongly disagree" and 3 representing "strongly agree."

SECONDARY OUTCOMES:
ACL-RSI questionnaire (Anterior Cruciate Ligament-Return to Sport after Injury) | One measurement during one visit at 4 to 24 months after surgery
  The ACL-RSI measures the patient's understanding of his knee. It comprises 12 questions with a score of 1 to 10 for each
Individual - age | One measurement during one visit at 4 to 24 months after surgery
  Personal characteristics recorded in the medical report as age
Strength | One measurement during one visit at 4 to 24 months after surgery
  Measurement of knee extensors and flexors peak strength (in newton.meter, Nm) on isokinetic dynamometer, part of the current Return-to-sport process
Surgery characteristics | One measurement during one visit at 4 to 24 months after surgery
  Surgery characteristics recorded in the medical report as the type of surgery,
IKDC Subjective Knee Evaluation | One measurement during one visit at 4 to 24 months after surgery
  The IKDC Subjective Knee Evaluation Form is scored by summing the individual item scores and converting the total to a scale of 0 to 100. Higher scores reflect better function and fewer symptoms, with the final score indicating overall knee function.
RISE-ACL scale for assessing Risk-taking Intention and Sport Engagement after ACL reconstruction for test-retest reliability | Two measurements at a 5-day interval
  A smaller sample of 28 participants will complete the scale twice, with a 5-day interval, to test its reproducibility. Scoring and minimum-maximum values will be defined at the development stage
Individual characteristics - gender | One measurement during one visit at 4 to 24 months after surgery
  Personal characteristics recorded in the medical report as gender
Individual characteristics - sport | One measurement during one visit at 4 to 24 months after surgery
  Personal characteristics recorded in the medical report as type of sport with sport level of practice
Individual characteristics - return to sport | One measurement during one visit at 4 to 24 months after surgery
  Personal characteristics recorded in the medical report as return to sport after the surgery

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Caen Normandy, Caen, Basse-Normandie, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Labrousse A, Reboursiere E, Remilly M, Roulland R, Mergenthaler G, Hulet C, Drigny J. Development and validation of a scale to assess risk-taking intentions during return to sport following anterior cruciate ligament reconstruction. J ISAKOS. 2025 Dec 18:101052. doi: 10.1016/j.jisako.2025.101052. Online ahead of print. PMID 41421604